CLINICAL TRIAL: NCT04064333
Title: Slow-Stream Expiratory Muscle Strength Training for Veterans With Dysphagia Living in Long-term Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI employment change
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Jessica Davenport, Speech-Language Pathologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Sunnybrook_Women'
Record Dates: First submitted 2019-08-16; First posted 2019-08-21 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Dysphagia, Oropharyngeal; Dysphagia; Dysphagia, Progressive; Aging; Aspiration Pneumonia; Cough
Keywords: EMST; RMST; Expiratory Muscle Strength Training; Respiratory Muscle Strength Training; Videofluoroscopy; Aspiration Pneumonia; Rehabilitation; Dysphagia; Cough; Geriatric; Aging; Older Adults
MeSH Terms: conditions — Deglutition Disorders; Pneumonia, Aspiration; Cough

STUDY DESIGN:
Intervention Model Description: This study will use an exploratory, cross sectional study design for the pre-post analysis of voluntary cough, measured through spirometry, laryngeal penetration/aspiration during swallow with thin liquids, measured under videofluoroscopy, and dysphagia-related quality of life, measured via questionnaire and diet texture modification scale. There is no control group; all participants will receive the same slow-stream expiratory muscle strength training protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Slow-Stream Expiratory Muscle Strength Training (Experimental): The therapy protocol consists of 12 sets of five breaths through the EMST150 device per week, in sessions of three or four sets (15 or 20 breaths). A typical schedule might be one 15 breath session four days per week, or one 20 breath session three days per week.
  Interventions: Device: Slow-Stream Expiratory Muscle Strength Training

INTERVENTIONS:
Device: Slow-Stream Expiratory Muscle Strength Training — All participants will receive an initial visit for training on the therapy protocol, use of a weekly therapy log to track breaths, and use and maintenance of the EMST device. This will constitute the first EMST session and will be included in the therapy log as Week 1, Day 1. Each participant will have a minimum of seven weekly check-in visits from the research assistant and/or a member of the research team, where the EMST150 resistance will be recorded and adjusted to maintain training at 75% of their maximum load, as measured using the EMST150 device instruction manual. During these check-in visits, participants will provide their completed weekly therapy log and receive a new log.
  Other Names: EMST150; Respiratory Muscle Strength Training; Expiratory Muscle Strength Training

SUMMARY:
Sunnybrook Veterans Centre (VC) is a long-term care (LTC) facility with many elderly residents living with swallowing disorders who are at high risk of developing pneumonia from aspirating food/liquid into their lungs. Expiratory muscle strength training (EMST) using a hand-held resistance device over a four week intensive program has been shown to have promising results in improving cough function and reducing aspiration during swallowing in older, community-dwelling adults. The purpose of this study is to explore whether a modified slow-stream protocol of EMST over eight weeks is an effective therapy for improving swallowing safety and lung clearance in elderly VC residents with swallowing disorders. Before and after the eight week therapy program, we will measure participants' cough under spirometry, swallowing under videofluoroscopy, and their swallowing-related quality of life and diet texture modification. A three month follow-up visit will measure swallowing-related quality of life again, as well as record incidence of respiratory tract infections requiring antibiotics in the last three months, to be compared with broader institutional data.

DETAILED DESCRIPTION:
This study will take place in Sunnybrook Veterans Centre (VC), a long-term care facility (LTC) with many residents above the age of 85 years living with dysphagia. These residents with dysphagia are at high risk of respiratory tract infections from aspiration of food/liquid particles into the lungs, exacerbated by factors like increased dependence for feeding and oral care, decreased mobility, multiple medical comorbidities, polypharmacy, and increased frailty.

Expiratory muscle strength training (EMST) applied within a four-week intensive program (25 sets/week) has had promising results in improving cough function and reducing laryngeal penetration/aspiration (P/A) during swallowing in community-dwelling adults above the age of 65 years. The EMST150 is a handheld device with adjustable resistance that trains respiratory muscles used in exhalation. One set is defined as five exhales through the device set at a resistance level of 75% of an individual's maximum load, with a one minute break between breaths.

The intensive four week EMST program outlined in previous literature was appropriate for the active, community-dwelling population they were studying. However, it would not be appropriate for most of the residents in the VC due to the extreme age, multiple medical comorbidities, increased frailty, and decreased functional independence in this population. An important aim of this study is to promote success by creating a protocol that fits into the average resident's schedule in a feasible way, but also has a similar number of total breaths through the device, in order to achieve clinical results. Resident perspective was sought from the Residents' Council executive and meeting attendees, and the final protocol was approved in a Residents' Council meeting. Participants would continue doing their usual therapies and activities with the EMST protocol being an add-on to that.

The purpose of this study is to explore whether a modified, slow-stream EMST protocol of 12 sets/week over eight weeks is an effective therapy for improving pulmonary clearance and swallowing safety in LTC residents above the age of 85 years who have dysphagia. Primary outcomes will be assessed through a pre-post analysis of voluntary cough strength measured using spirometry, as well as laryngeal P/A measured under videofluoroscopy. Secondary outcome of swallowing-related quality of life will be measured using Dysphagia Handicap Index - Emotional scale and the International Dysphagia Diet Standardization Initiative Functional Diet Scale pre and post intervention, as well as at a 3 month follow-up. Incidence of respiratory tract infections requiring antibiotics in the three months post-intervention will be measured and compared with broader institutional data.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in the English language
* Identified by their speech-language pathologist as at risk for laryngeal penetration/aspiration when drinking thin liquids
* A Penetration Aspiration Scale score of 3+ on at least one thin liquid bolus during pre-test videofluoroscopy, as rated live at the time of test by the speech-language pathologist conducting the videofluoroscopy.
* Cognitively and physically able to perform study tasks (spirometry, EMST). If assistance and/or cuing is required, the participant must have a support team who is agreeable to providing this for the duration of the study at time of consent. Support teams may consist of any combination of family, friends, private companions, and VC staff.
* Medical clearance by the participant's most responsible physician (MRP)

Exclusion Criteria:

At time of consent

* General medical exclusions: Any history of hernia, pneumothorax, perforated tympanic membrane, recent surgery, untreated gastroesophageal reflux disease or untreated hypertension.
* Other medical conditions where increased intrathoracic pressure would be contraindicated, on an individual basis, as per participant's MRP
* Cognitively and/or physically unable to perform study tasks, despite support
* Participants who do not consent to videofluoroscopy or for whom videofluoroscopy is contraindicated

After time of consent

* Participants who score PAS < 3 on pre-test videofluoroscopy
* Inability to complete pre-post testing for at least one primary outcome
* Inability to complete minimum 50 breaths of the weekly protocol, and minimum 400 total breaths through the device over the 8 week program

Ages: 85 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Voluntary Cough Volume Acceleration | Pre-treatment baseline, 10 weeks after baseline
  Change in maximum voluntary cough strength pre and post intervention as measured through airflow analysis of digital cough waveform.
  The digital waveform will provide measures of inspiratory phase duration (seconds), compression phase duration (seconds), expiratory rise time (seconds), and expiratory peak flow (Litres/second), and cough volume acceleration (Litres/second squared) will be calculated as expiratory peak flow/expiratory phase rise time, as in Pitts et al., 2019, to represent cough strength.
  The protocol will consist of three voluntary coughs into a spirometer using a nose-clip, with a brief rest of 30-60 seconds between attempts. The best effort will be used to generate a digital cough waveform to be analyzed separately by two trained raters consisting of members of the research team or research assistant. Any disagreements between raters will be resolved through consensus with a third rater.
Penetration Aspiration Scale (PAS) | Pre-treatment baseline, 10 weeks after baseline
  Change in frequency of laryngeal penetration (PAS scores >2) and aspiration (PAS scores >5) on swallows of thin liquid pre and post intervention.
  Videofluoroscopy (VFSS) protocol of four 10 mL thin liquid consisting of 20% w/v concentration of barium (Polibar Plus) and water, performed by the speech-language pathologist (SLP). Video processing will include removing audio, splicing the recordings into deidentified bolus-length clips, and randomizing these for rating. These clips will be rated using the Penetration Aspiration Scale by three SLPs who will attend calibration training at the Swallowing Rehabilitation Research Laboratory at Toronto Rehabilitation Institute. Raters will be blinded to participant and time. All raters will overlap on the first 25 clips, from which inter-rater reliability measures will be taken, and with any disagreements being resolved through consensus. The remaining clips will be divided among the three raters.

SECONDARY OUTCOMES:
Dysphagia Handicap Index Emotional Subscale (DysHI-E) | Pre-treatment baseline, 10 weeks after baseline, 3 months post-intervention
  Change in swallowing-related quality of life. The DysHI-E consists of seven questions answered using a 3-point scale of Never, Sometimes, and Always, and a 7-point severity scale ranging from 1-normal to 7-severe problem (Silbergleit et al., 2012). This will be converted into a visual analogue scale and responses will be measured in centimeters from left to right, with the far left end being Never or 0.00 cm, and the far right end being Always or 30.00 cm.
International Dysphagia Diet Standardization Initiative Functional Diet Scale (IDDSI-FDS) | Pre-treatment baseline, 10 weeks after baseline, 3 months post-intervention
  Change in the level of diet texture restriction secondary to dysphagia. The IDDSI-FDS measures the number of diet texture levels allowed from the International Dysphagia Diet Standardization Initiative Framework.

OTHER OUTCOMES:
Incidence of Respiratory Tract Infections Requiring Antibiotics | 3 months post-intervention
  Incidence of respiratory tract infections requiring antibiotics over the three months following intervention, for comparison with broader institutional data.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa DiProspero, MRT BSc MSc, Study Director — Director, Practice-Based Research and Innovation; Jessica Davenport, MHSc, S-LP, Principal Investigator — Speech-Language Pathologist, Sunnybrook
Locations (1):
- Sunnybrook Health Sciences Centre - Veterans Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] Bonilha HS, Huda W, Wilmskoetter J, Martin-Harris B, Tipnis SV. Radiation Risks to Adult Patients Undergoing Modified Barium Swallow Studies. Dysphagia. 2019 Dec;34(6):922-929. doi: 10.1007/s00455-019-09993-w. Epub 2019 Mar 4. PMID 30830303
- [Background] Kim J, Davenport P, Sapienza C. Effect of expiratory muscle strength training on elderly cough function. Arch Gerontol Geriatr. 2009 May-Jun;48(3):361-6. doi: 10.1016/j.archger.2008.03.006. Epub 2008 May 23. PMID 18457885
- [Background] Tada A, Matsumoto H, Soda R, Endo S, Kawai H, Kimura G, Yamashita M, Okada C, Takahashi K. [Effects of pulmonary rehabilitation in patients with pulmonary tuberculosis sequelae]. Nihon Kokyuki Gakkai Zasshi. 2002 Apr;40(4):275-81. Japanese. PMID 12096494
- [Background] Park JS, Oh DH, Chang MY. Effect of expiratory muscle strength training on swallowing-related muscle strength in community-dwelling elderly individuals: a randomized controlled trial. Gerodontology. 2017 Mar;34(1):121-128. doi: 10.1111/ger.12234. Epub 2016 May 16. PMID 27198586
- [Background] Pitts T, Bolser D, Rosenbek J, Troche M, Okun MS, Sapienza C. Impact of expiratory muscle strength training on voluntary cough and swallow function in Parkinson disease. Chest. 2009 May;135(5):1301-1308. doi: 10.1378/chest.08-1389. Epub 2008 Nov 24. PMID 19029430
- [Background] Silbergleit AK, Schultz L, Jacobson BH, Beardsley T, Johnson AF. The Dysphagia handicap index: development and validation. Dysphagia. 2012 Mar;27(1):46-52. doi: 10.1007/s00455-011-9336-2. Epub 2011 Mar 20. PMID 21424584
- [Background] Steele CM, Grace-Martin K. Reflections on Clinical and Statistical Use of the Penetration-Aspiration Scale. Dysphagia. 2017 Oct;32(5):601-616. doi: 10.1007/s00455-017-9809-z. Epub 2017 May 22. PMID 28534064
- [Background] Stokely SL, Molfenter SM, Steele CM. Effects of barium concentration on oropharyngeal swallow timing measures. Dysphagia. 2014 Feb;29(1):78-82. doi: 10.1007/s00455-013-9485-6. Epub 2013 Sep 18. PMID 24045851
- [Background] Troche MS, Okun MS, Rosenbek JC, Musson N, Fernandez HH, Rodriguez R, Romrell J, Pitts T, Wheeler-Hegland KM, Sapienza CM. Aspiration and swallowing in Parkinson disease and rehabilitation with EMST: a randomized trial. Neurology. 2010 Nov 23;75(21):1912-9. doi: 10.1212/WNL.0b013e3181fef115. PMID 21098406
- [Background] Weening-Dijksterhuis E, de Greef MH, Scherder EJ, Slaets JP, van der Schans CP. Frail institutionalized older persons: A comprehensive review on physical exercise, physical fitness, activities of daily living, and quality-of-life. Am J Phys Med Rehabil. 2011 Feb;90(2):156-68. doi: 10.1097/PHM.0b013e3181f703ef. PMID 20881587
- [Background] Leung G, Katz PR, Karuza J, Arling GW, Chan A, Berall A, Fallah S, Binns MA, Naglie G. Slow Stream Rehabilitation: A New Model of Post-Acute Care. J Am Med Dir Assoc. 2016 Mar 1;17(3):238-43. doi: 10.1016/j.jamda.2015.10.016. Epub 2015 Dec 2. PMID 26654839
- [Background] Steele CM, Namasivayam-MacDonald AM, Guida BT, Cichero JA, Duivestein J, Hanson B, Lam P, Riquelme LF. Creation and Initial Validation of the International Dysphagia Diet Standardisation Initiative Functional Diet Scale. Arch Phys Med Rehabil. 2018 May;99(5):934-944. doi: 10.1016/j.apmr.2018.01.012. Epub 2018 Feb 8. PMID 29428348
- See also: Website of Expiratory Muscle Strength Trainer (EMST150) used in protocol — http://emst150.com/
- See also: Website of International Dysphagia Diet Standardization Initiative, basis of Functional Diet Scale — http://iddsi.org/